CLINICAL TRIAL: NCT06766253
Title: The Effects of GMA-TULIP, I-gel, and BlockBuster Laryngeal Mask in Laparoscopic Surgeries With Trendelenburg Position Under General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.135
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-07

CONDITIONS: Sore-throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GMA-TULIP (Experimental): Using GMA-TULIP non-inflatable laryngeal mask for airway management in patients who receives laparoscopic surgeries with trendelenburg position.
  Interventions: Device: GMA-TULIP
- i-gel (Active Comparator): Using i-gel non-inflatable laryngeal mask for airway management in patients who receives laparoscopic surgeries with trendelenburg position.
  Interventions: Device: GMA-TULIP
- BlockBuster (Active Comparator): Using BlockBuster inflatable laryngeal mask for airway management in patients who receives laparoscopic surgeries with trendelenburg position.
  Interventions: Device: GMA-TULIP

INTERVENTIONS:
Device: GMA-TULIP — Using GMA-TULIP non-inflatable laryngeal mask for airway management in patients who receives laparoscopic surgeries with trendelenburg position.

SUMMARY:
This project aims to compare the application effects of traditional inflatable BlockBuster laryngeal mask, i-gel non-inflatable laryngeal mask and GMA-TULIP non-inflatable laryngeal mask in laparoscopic surgeries with trendelenburg position under general anesthesia, in order to explore which laryngeal mask is best for reducing postoperative throat pain of patients and improving patient comfort and satisfaction.

DETAILED DESCRIPTION:
Laryngeal mask and tracheal intubation are the two most commonly used airway management methods for patients under general anesthesia. Compared with tracheal intubation, laryngeal mask has the advantages of simple insertion, less airway injury, and more stable hemodynamics. Therefore, laryngeal mask has been widely used in airway management during general anesthesia. Studies have shown that about 3 million patients in the British National Health Service system receive anesthesia surgery with different types of airway management every year, and the usage rate of laryngeal mask is higher than that of tracheal intubation, accounting for about 56.2%.

Many new laryngeal masks have been improved based on the classic laryngeal mask and applied to clinical practice. Currently, there are two main types of laryngeal masks: inflatable laryngeal masks and non-inflatable laryngeal masks. Inflatable laryngeal masks are traditional types, including BlockBuster, Superme, ProSeal, and Fastrach, which are the most widely used in clinical practice. Traditional laryngeal masks require inflation to achieve sealing of the throat opening, but inflatable laryngeal masks have drawbacks such as inconvenient insertion, higher incidence of oral and pharyngeal injury and bleeding, and a higher incidence of postoperative sore throat. According to report, the incidence of postoperative sore throat with laryngeal masks is up to 31.9%.

The non-inflatable laryngeal mask is mirrored at the throat opening and made of thermoplastic elastomer material, which achieves a gas tightness effect similar to the inflatable laryngeal mask, improves the ease of insertion, and reduces complications such as sore throat and mucosal injury and bleeding. The i-gel laryngeal mask is the most commonly used non-inflated laryngeal mask currently. A meta-analysis found that the incidence of postoperative sore throat with the i-gel laryngeal mask is 4.1%, which is significantly lower than that of inflatable laryngeal masks.

GMA-TULIP is a new type of non-inflatable laryngeal mask with advantages such as C-shaped double gastric tube channel, stable platform for tongue root, soft tissue sealing ring, epiglottis attached protrusion, and consistent with the anatomical structure of the throat. In addition, the front cuff of GMA-TULIP is small, which only needs to reach the two sides of the pyriform fossa in the distal end. During placement, it passes over the tongue root and reaches the standard position. Compared with i-gel non-inflatable laryngeal mask, GMA-TULIP is more in line with the anatomical position design, theoretically better in position, less likely to cause damage to the throat and pharynx, thus, lower incidence of postoperative sore throat.

In laparoscopic surgeries with trendelenburg position under general anesthesia, the airway pressure is significantly higher than that in the supine position and non-laparoscopic surgery, thus, the incidence of postoperative sore throat is higher than that in the supine position and non-laparoscopic surgery. Therefore, this project intends to compare the effects of traditional inflatable BlockBuster laryngeal mask, i-gel non-inflatable laryngeal mask, and GMA-TULIP non-inflatable laryngeal mask in laparoscopic surgeries with trendelenburg position, in order to explore which laryngeal mask is best for reducing postoperative throat pain of patients and improving patient comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients received laparoscopic surgeries with trendelenburg position and an estimated surgery duration of less than 3 hours.
2. Ages between 18 to 80, and body mass index less than 28 kg/m².
3. American Society of Anesthesiologists (ASA) Grades I-III.
4. Patients are willing to participate and be able to understand and sign an informed consent form.

Exclusion Criteria:

1. Patients with a mouth opening less than 2 cm.
2. Patients with risk factors for regurgitation and aspiration of gastric contents.
3. Patients with laryngopharyngeal diseases.
4. Patients with potentially difficult airways.
5. Patients with hearing, intellectual, communication, and cognitive impairments.
6. Any reason that patients could not cooperate with the study or that the researcher deems inappropriate for inclusion in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat | 10 minutes, 2 hours, 24 hours, 48 hours, and 72 hours after surgery
  Sore throat is assessed by Prince-Henry pain scores (0 to 4 points)

SECONDARY OUTCOMES:
incidence of dysphagia | 10 minutes, 2 hours, 24 hours, 48 hours, and 72 hours after surgery
  Check the patient can swallow or not

OTHER OUTCOMES:
Time of insertion | 1 min after successful insertion of the laryngeal mask
  Insertion time was defined as the time from the opening of the mouth by the operator to the positively insert the laryngeal mask. The time of glottic examination, adjustment between two ventilation insertions, and ventilation was not measured as ventilation insertion time.
Times of laryngeal mask adjustment before the successful insertion | 1 min after the airway is successfully controlled.
  The times of laryngeal mask adjustments before successful laryngeal mask insertion.
The rate of first-insertion success | 1 min after the first-attempt insertion of the laryngeal mask
  The first successful insertion is defined as oropharyngeal leak pressure higher than 20 cmH2O and grade 1-2 of the laryngeal view under the fibreoptic bronchoscopy (indicating the accuracy of laryngeal mask positioning) at the first attempt.
Total insertion success rate | 1 min after the airway is successfully controlled.
  The total successful insertion is defined as ventilation with the allocated laryngeal mask after anesthesia induction.
Success rate of gastric tube insertion through laryngeal mask | 1 min after the laryngeal mask is successful inserted
  After the laryngeal mask is successful inserted, a fully lubricated 14F gastric tube was inserted through its esophageal drainage tube
grade of view on fibreoptic bronchoscopy | 1 min after successful insertion of the laryngeal mask, 5 min after pneumoperitoneum and trendelenburg position
  After successful insertion of the laryngeal mask, fiberoptic bronchoscopy was used and graded according to the degree of glottic and epiglottis exposure by a 4-point scale system: 1, full view of glottis; 2, vocal cords, arytenoids, and inferior surface of epiglottis visible; 3, only superior surface of epiglottis visible; 4, no part of epiglottis or larynx visible. The grades 1 and 2 were defined as optimal fiberscopic view.
oropharyngeal leak pressure | 1 min after the laryngeal mask is successfully inserted, 5 min after pneumoperitoneum and trendelenburg position
  After the laryngeal mask is inserted, set the fresh gas flow to 3 L/min in manual mode, turn the APL valve to 30 cmH2O, and listen to the neck until the sound of air leakage is heard. The peak airway pressure at this time is the oropharyngeal leak pressure.
Peak airway pressure | 1 min after the laryngeal mask is successfully inserted, 5 min after pneumoperitoneum and trendelenburg position
  Peak pressure refers to the maximum pressure produced by the airflow in the closed circuit each time the ventilator delivers a certain amount of gas from the endotracheal tube to the patient's lungs. Peak airway pressure was measured by the anesthesia machine automatically.
Airway plateau pressure | 1 min after the laryngeal mask is successfully inserted, 5 min after pneumoperitoneum and trendelenburg position
  Plateau airway pressure refers to the pressure that a certain amount of gas remains in the lungs against the entire closed system at the end of the passage of air, before the beginning of exhalation. Airway plateau pressure was measured by the anesthesia machine automatically.
heart rate | 1 min before laryngeal mask insertion or withdrawn, and 1 min after the laryngeal mask is inserted or withdrawn
  heart rate
diastolic blood pressure | 1 min before laryngeal mask insertion or withdrawn, and 1 min after the laryngeal mask is inserted or withdrawn
  diastolic blood pressure
systolic blood pressure | 1 min before laryngeal mask insertion or withdrawn, and 1 min after the laryngeal mask is inserted or withdrawn
  systolic blood pressure
mean arterial pressure | 1 min before laryngeal mask insertion or withdrawn, and 1 min after the laryngeal mask is inserted or withdrawn
  mean arterial pressure
Times of intraoperative air leakage | From the start of anesthesia to the end of the anesthesia
  intraoperative air leakage is defined as hearing an air leak in the pharynx during the operation
Times of laryngeal mask adjustment during the operation | From the start of anesthesia to the patient's exit from the operating room
  the times of the laryngeal mask adjustment during the operation were recorded
The incidence of aspiration | From the start of anesthesia to the patient's exit from the operating room
  The aspiration is defined as seeing the gastric content in the trachea
The incidence of regurgitation | From the start of anesthesia to the patient's exit from the operating room
  The regurgitation is defined as seeing the gastric content in the mouth
incidence of blood staining on the laryngeal mask | 1 min after the laryngeal mask is pull out after surgery.
  When the laryngeal mask was pulled out, the laryngeal mask was stained with blood
The incidence of cough | the time when the laryngeal mask is pull out
  When the laryngeal mask was pulled out, record whether the patient has cough or not.
Active mouth bleeding rate | 1 min after laryngeal mask removal
  After the laryngeal mask was removed, record whether active bleeding occurred at the patient's mouth
Time of laryngeal mask application | 1 min after the laryngeal mask is withdrawn
  The time of laryngeal mask withdrawn minus the time of successful laryngeal mask insertion is the time of laryngeal mask application
Length of surgery | 1 min after the end of surgery
  The end of the surgery time minus the start of the surgery time is the length of surgery
The incidence of hoarseness | 10 minutes, 2 hours, 24 hours, 48 hours, and 72 hours after surgery
  the patient is hoarse when speaking

CONTACTS AND LOCATIONS:
Overall Officials: Bing Chen, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available with the responding author when required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available when publish and keep it for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal.